CLINICAL TRIAL: NCT04902196
Title: Acute Effects of a High Intensity Training Protocol on Pain Processing and Inflammatory Parameters in Persons With Chronic Nonspecific Low Back Pain.
Brief Title: Acute Effects of High Intensity Training on Pain Processing and Inflammation in Chronic Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Annick Timmermans, Principal Investigator, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPB-QST-001
Record Dates: First submitted 2021-05-07; First posted 2021-05-26 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Low Back Pain; Inflammation
MeSH Terms: conditions — Low Back Pain; Inflammation

STUDY DESIGN:
Intervention Model Description: group 1: 2 testmoments, min. 7 days and max. 14 days in between them. Both have exactly the same design and the same content of measurements, with the exception of the intensity of the performed exercise protocol. The correct wattage for the exercise protocols is extracted from a previous maximum exercise test at the Jessa Hospital. By means of a randomized cross-over design, participants from group 1 will undergo both a moderately intensive cardiorespiratory protocol (MIT) and a high-intensity cardiorespiratory protocol (HIT).
  group 2: 2 testmoments, min. 7 days and max. 14 days in between them. During the first testmoment, a maximum exercise test is performed (to establish the exercise protocol that will be used during the second testmoment). The design and content of the second test moment is identical to that of group 1 with the exception of 1) only performing a HIT protocol and 2) not completing the questionnaires only applicable for persons with low back pain (i.e. ODI, BPI).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): persons with chronic low back pain of an non-specific origin
  Interventions: Other: high intensity cardiorespiratory exercise protocol; Other: moderate intensity cardiorespiratory exercise protocol
- Group 2 (Control group) (Active Comparator): "healthy" persons (pain-free)
  Interventions: Other: high intensity cardiorespiratory exercise protocol

INTERVENTIONS:
Other: high intensity cardiorespiratory exercise protocol — During the high intensive cardiorespiratory exercise protocol, a bicycle ergometer (eBike Basic, General Electric GmbH, Bitz, Germany) with pulmonary gas exchange analysis (MetaMax 3B, Cortex Biophysik GmbH, Leipzig, Germany) will be used. Oxygen uptake (VO2max), expiratory volume (VE) and respiratory exchange rate (RER) will be tracked every breath and an average will be taken every 10s. Heart rate is continuously monitored using a heart rate chest strap (Polar Electro Inc., Finland). After a five-minute warm-up, a high-intensity interval protocol is started, consisting of five one-minute bouts (110 reps/minute at 100% VO2max workload), separated by one minute of active rest (75 reps per minute at 50% VO2max workload).
  Other Names: physical perfomance intervention
Other: moderate intensity cardiorespiratory exercise protocol — During the moderate intensive cardiorespiratory exercise protocol, a bicycle ergometer (eBike Basic, General Electric GmbH, Bitz, Germany) with pulmonary gas exchange analysis (MetaMax 3B, Cortex Biophysik GmbH, Leipzig, Germany) will be used. Oxygen uptake (VO2max), expiratory volume (VE) and respiratory exchange rate (RER) will be tracked every breath and an average will be taken every 10s. Heart rate is continuously monitored using a heart rate chest strap (Polar Electro Inc., Finland). After a five-minute warm-up, participants begin a moderately-intensive continuous 14-minute exercise protocol at a stable resistance (90 repetitions per minute at 60% VO2max workload).
  Other Names: physical perfomance intervention
  Arms: Group 1

SUMMARY:
A multitude of exercise therapy modalities are effective in improving daily physical function and relieving pain in various forms of chronic musculoskeletal pain (CMP) such as chronic neck pain, osteoarthritis, fibromyalgia, and chronic low back pain. However, the inital pain response to physical exercise can be variable in populations with CMP. Indeed, some studies show no change or even brief exacerbations in pain in individuals with CMP in response to exercise. These pain flare-ups in chronic pain populations are believed to be associated with increased pain sensitivity after exercise.

The magnitude of "exercise-induced hypoalgesia" or the EIH response (i.e., the short-term endogenous pain-suppressing response after exercise) is believed to depend on several training factors, including exercise intensity. Currently, there is limited understanding of the optimal intensity of exercise for producing hypoalgesic effects on different types of pain stimuli. Nevertheless, several indications have been found for a dose-response effect in exercise and the amount of EIH that can be expected. However, very few studies have specifically examined EIH in people with chronic low back pain, although exercise is recommended in national and international guidelines as a basic treatment for the treatment of this condition.

Relevant studies have also shown that exercise can induce an extensive inflammatory response in CMP, which may contribute to the disrupted EIH production. In addition, it is stated that this inflammatory response in CMP is also influenced by psychosocial factors.

Therefore, the aim of the current cross-sectional cohort study is to expand the knowledge of the pain processing and inflammatory response to acute physical exertion in persons with chronic low back pain through evaluation responses of persons with this disorder to a high intensity training protocol. It is also investigated whether their EIH response is dependent on psychosocial factors.

DETAILED DESCRIPTION:
Chronic musculoskeletal pain (CMP) currently affects up to 20% of all people or about 1.5 billion persons worldwide, and these numbers continue to increase steadily. CMP can have a significant impact on both the physical and psychological functioning of an individual with consequences including recurring health care costs, limitation of participation in society, and long-term absenteeism. This makes CMP a pervasive medical problem that consumes a huge amount of healthcare resources.

Regular physical activity and exercise can impact many aspects of a person's general health through improving both physical functioning (e.g. cardiorespiratory fitness), as well as psychological functioning (e.g. mental health). Moreover, many common forms of exercise therapy have been studied and shown to be effective in relieving pain. These include amongst others running, walking, resistance training, water training and Tai Chi. As a result, more and more studies are referring to exercise therapy as an accessible, cost-effective and cost-effective therapeutic modality for the treatment of almost all types of musculoskeletal disorders. For example, substantial evidence already supports that exercise therapy can be effective in improving daily physical function and relieving pain in individuals with chronic neck pain, osteoarthritis, fibromyalgia and chronic low back pain.

While exercise therapy thus has clear benefits in persons with CMP, pain response to exercise can be variable in these populations, especially in the initial stages of therapy. Indeed, some studies show no change or even brief exacerbations of pain in persons with CMP in response to exercise. These 'flare-ups' of acute pain during exercise are believed to be related to increased chronic pain sensitivity.

The effect of "exercise-induced hypoalgesia" or EIH (i.e., the short-term endogenous pain-inhibiting response after exercise) is well documented in healthy subjects. The magnitude of the EIH response is believed to depend on several factors, including the type, dose, and intensity of the exercise. While the EIH response, measured as a change in the pain threshold after exercise, can be assess with quantitative sensory tests (ie a panel of diagnostic tests used to assess somatosensory function), there is currently only limited understanding of the optimal exercise intensity to produce hypoalgesic effects on different types of pain stimuli. Nevertheless, several indications of a dose-response effect in exercise and the amount of EIH that can be expected have been found. Studies have also shown that EIH can be affected in a variety of musculoskeletal pain disorders, including whiplash, knee osteoarthritis, or shoulder pain. This may explain the varied response to exercise and may have important implications for exercise prescription. However, very few studies have examined the relationship between exercise modalities and EIH in people with chronic low back pain, although exercise is recommended in national and international guidelines as a basic treatment for the treatment of this condition.

Furthermore, research has also shown that exercise can induce an extensive inflammatory response in persons with CMP (by drastically changing levels of inflammatory markers at various sites in the nervous system), which may heavily contribute to the disrupted production of EIH. Specifically, the effect of interleukin-6 (IL-6) during physical performance as a potential local "pain trigger" is gaining more and more attention. Recently, several pathological pain models have shown significantly increased expression levels of IL-6 and its receptor in the spinal cord and dorsal root ganglia.

In addition, these inflammatory responses and EIH are said to be influenced by psychosocial factors in chronic pain disorders. For example, higher anxiety and catastrophe resulted in an enhanced pro-inflammatory response in fibromyalgia and osteoarthritis. Likewise, sleep disturbances resulted in higher IL-6 levels in CLBP. As such, these results suggest that EIH can be affected by multiple cellular and molecular events in the pain process as well as individual responses to specific situations.

The objective of this study is to expand the knowledge of the pain processing and inflammatory response to acute physical exertion of persons with chronic low back pain. This study will also investigate whether these responses are dependent on psychosocial factors. The information provided by this study may contribute to a better understanding of the mechanisms that lead to varied responses to exercise in people with chronic low back pain. This allows therapy protocols to be adapted and the worsening of symptoms in some people with chronic low back pain to be counteracted by these therapy protocols.

Primary research questions:

* Question 1: To what extent does a single high or moderately intensive cardiorespiratory exercise protocol have an acute effect on pain processing and the inflammatory response in persons with chronic low back pain?
* Question 2: To what extent is the acute effect of a single high or moderately intensive cardiorespiratory exercise protocol on pain processing and the inflammatory response correlated with differences in psychosocial parameters in persons with chronic low back pain?
* Question 3: To what extent is the acute effect of a single high or moderately intensive cardiorespiratory exercise protocol on pain processing and the inflammatory response in subjects with chronic low back pain different from healthy subjects?

ELIGIBILITY:
Inclusion criteria for group 1 (persons with chronic low back pain)

* Primary complaint: non-specific chronic low back pain.

  * Low back pain is defined as pain in the area between the lower ribs and the upper buttock crease, with or without radiation in the leg
  * Chronic: current episode > 12 weeks, mean pain intensity between 3-8/10
  * Non-specific: the main pain cannot be traced back to a known pathology
* Age: 18-65 years
* Acute pain intensity at the time of testing between 3-8/10 (i.e. a pain intensity within this range is necessary to obtain a correct estimate of the pain response)
* Understanding of the Dutch language (written and spoken)

Inclusion criteria for group 2 (healthy persons)

* No acute or chronic musculoskeletal complaints (i.e. VAS> 2/10 in the last 24 hours)
* Age: 18-65 years
* Understanding of the Dutch language (written and spoken)

Exclusion criteria for both group 1 and 2

* Invasive spinal surgery within the last 18 months (arthrodesis will always be excluded, microsurgery is allowed)
* Radiculopathy (uni- or bilateral) of the lower extremities
* Comorbidities: paresis and sensory disturbances with a neurological cause in the lower extremities, diabetes mellitus, rheumatoid arthritis, autoimmune disorders etc.
* Pregnancy
* Ongoing compensation complaints and/or incapacity for work > 6 months
* Previous active rehabilitation (i.e. exercise therapy) for low back pain in the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
blood sample (evaluation of inflammatory markers) - IL-6 concentration | baseline
  Two venous blood sample (serum) will be collected (one blood sample before the first QST protocol and one after the cardiorespiratory exercise protocol) by venous puncture. All samples are kept at room temperature for two hours. Afterwards, they are centrifuged at 1300 g for 15 minutes, transferred to cryovials (4 cryovials of 500µl), and stored at -80 ° C in the University Biobank Limburg (UBiLim) until further processing and analysis. Inflammatory markers will be assayed via bead-based multiplex assay using flow cytometry i.e. LegendPlex Multiplex Assay, inflammation panel 1. Absorbance is measured with an automated Microplate Reader.
  With this panel plasma IL-6 concentration (pg/ml) will be evaluated.
blood sample (evaluation of inflammatory markers) - TNF-α concentration | baseline
  Two venous blood sample (serum) will be collected (one blood sample before the first QST protocol and one after the cardiorespiratory exercise protocol) by venous puncture. All samples are kept at room temperature for two hours. Afterwards, they are centrifuged at 1300 g for 15 minutes, transferred to cryovials (4 cryovials of 500µl), and stored at -80 ° C in the University Biobank Limburg (UBiLim) until further processing and analysis. Inflammatory markers will be assayed via bead-based multiplex assay using flow cytometry i.e. LegendPlex Multiplex Assay, inflammation panel 1. Absorbance is measured with an automated Microplate Reader.
  With this panel plasma TNF-α concentration (pg/ml) will be evaluated.
blood sample (evaluation of inflammatory markers) - IL-6 concentration | Day 7
  Two venous blood sample (serum) will be collected (one blood sample before the first QST protocol and one after the cardiorespiratory exercise protocol) by venous puncture. All samples are kept at room temperature for two hours. Afterwards, they are centrifuged at 1300 g for 15 minutes, transferred to cryovials (4 cryovials of 500µl), and stored at -80 ° C in the University Biobank Limburg (UBiLim) until further processing and analysis. Inflammatory markers will be assayed via bead-based multiplex assay using flow cytometry i.e. LegendPlex Multiplex Assay, inflammation panel 1. Absorbance is measured with an automated Microplate Reader.
  With this panel plasma IL-6 concentration (pg/ml) will be evaluated.
blood sample (evaluation of inflammatory markers) - TNF-α concentration | Day 7
  Two venous blood sample (serum) will be collected (one blood sample before the first QST protocol and one after the cardiorespiratory exercise protocol) by venous puncture. All samples are kept at room temperature for two hours. Afterwards, they are centrifuged at 1300 g for 15 minutes, transferred to cryovials (4 cryovials of 500µl), and stored at -80 ° C in the University Biobank Limburg (UBiLim) until further processing and analysis. Inflammatory markers will be assayed via bead-based multiplex assay using flow cytometry i.e. LegendPlex Multiplex Assay, inflammation panel 1. Absorbance is measured with an automated Microplate Reader.
  With this panel plasma TNF-α concentration (pg/ml) will be evaluated.
QST protocol (evaluation of pain processing) - local pressure pain thresholds | Baseline
  Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing before and after the cardiorespiratory exercise protocol. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. A standardized 20-minute test protocol serves as the basis.
  Two local pressure pain thresholds scores, displayed as kilogram-force (or KgF), 1 at the left and 1 at the right level of the lower back (at the subjective pain level) will be determined using a manual algometer (Force Ten FDX 50; Wagner Instruments, Greenwich, CT). Pressure will be applied at a constant rate of approximately 1 kg/s. Measurements at each side are performed twice with 5 minutes of rest apart. The highest score is used for analysis.
QST protocol (evaluation of pain processing) - widespread mechanical hyperalgesia | Baseline
  Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing before and after the cardiorespiratory exercise protocol. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. A standardized 20-minute test protocol serves as the basis.
  Widespread mechanical hyperalgesia (1 protocol, 3 scores for each leg displayed in Newton) will be measured by determining the Cuff pressure pain threshold (cPPT), cuff pressure pain tolerance (cPTT), and cuff pressure pain tolerance limit (cPTL) during increased cuff pressure with a rate of 1 kPa/s by a computer-controlled cuff pressure algometer (NociTech, Denmark, and Aalborg University, Denmark) at the level of the left and right leg (calve).
QST protocol (evaluation of pain processing) - temporal summation | Baseline
  Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing before and after the cardiorespiratory exercise protocol. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. A standardized 20-minute test protocol serves as the basis.
  Temporal summation of pain (1 protocol, 10 scores displayed in Newton) will be measured by determining pressure pain thresholds during 10 repeated cuff pressure stimulations (2-second duration and 1-second interval between stimuli) by a computer-controlled cuff pressure algometer (NociTech, Denmark, and Aalborg University, Denmark) at the level of the dominant leg (calve).
QST protocol (evaluation of pain processing) - conditioned pain modulation | Baseline
  Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing before and after the cardiorespiratory exercise protocol. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. A standardized 20-minute test protocol serves as the basis.
  Conditioned pain modulation ('CPM', 1 protocol, 3 scores for the dominant leg displayed in Newton) will be explored to evaluate the endogenous analgesic system by examining the change in the Cuff pressure pain threshold (cPPT), cuff pressure pain tolerance (cPTT), and cuff pressure pain tolerance limit (cPTL) seen in one body area ('test stimulus') due to pain induced in another body area ('conditioned stimulus') by a computer-controlled cuff pressure algometer (NociTech, Denmark, and Aalborg University, Denmark) at the level of the dominant leg (calve) for the test stimulus and the non-dominant leg for the conditioning stimulus.
QST protocol (evaluation of pain processing) - local pressure pain thresholds | day 7
  Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing before and after the cardiorespiratory exercise protocol. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. A standardized 20-minute test protocol serves as the basis.
  Two local pressure pain thresholds scores, displayed as kilogram-force (or KgF), 1 at the left and 1 at the right level of the lower back (at the subjective pain level) will be determined using a manual algometer (Force Ten FDX 50; Wagner Instruments, Greenwich, CT). Pressure will be applied at a constant rate of approximately 1 kg/s. Measurements at each side are performed twice with 5 minutes of rest apart. The highest score is used for analysis.
QST protocol (evaluation of pain processing) - widespread mechanical hyperalgesia | day 7
  Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing before and after the cardiorespiratory exercise protocol. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. A standardized 20-minute test protocol serves as the basis.
  Widespread mechanical hyperalgesia (1 protocol, 3 scores for each leg displayed in Newton) will be measured by determining the Cuff pressure pain threshold (cPPT), cuff pressure pain tolerance (cPTT), and cuff pressure pain tolerance limit (cPTL) during increased cuff pressure with a rate of 1 kPa/s by a computer-controlled cuff pressure algometer (NociTech, Denmark, and Aalborg University, Denmark) at the level of the left and right leg (calve).
QST protocol (evaluation of pain processing) - temporal summation | day 7
  Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing before and after the cardiorespiratory exercise protocol. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. A standardized 20-minute test protocol serves as the basis.
  Temporal summation of pain (1 protocol, 10 scores displayed in Newton) will be measured by determining pressure pain thresholds during 10 repeated cuff pressure stimulations (2-second duration and 1-second interval between stimuli) by a computer-controlled cuff pressure algometer (NociTech, Denmark, and Aalborg University, Denmark) at the level of the dominant leg (calve).
QST protocol (evaluation of pain processing) - conditioned pain modulation | day 7
  Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing before and after the cardiorespiratory exercise protocol. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. A standardized 20-minute test protocol serves as the basis.
  Conditioned pain modulation ('CPM', 1 protocol, 3 scores for the dominant leg displayed in Newton) will be explored to evaluate the endogenous analgesic system by examining the change in the Cuff pressure pain threshold (cPPT), cuff pressure pain tolerance (cPTT), and cuff pressure pain tolerance limit (cPTL) seen in one body area ('test stimulus') due to pain induced in another body area ('conditioned stimulus') by a computer-controlled cuff pressure algometer (NociTech, Denmark, and Aalborg University, Denmark) at the level of the dominant leg (calve) for the test stimulus and the non-dominant leg for the conditioning stimulus.

SECONDARY OUTCOMES:
The Brief Pain Inventory short form (BPI-sf) | Baseline
  This nine-item questionnaire is used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The patient is asked to rate the worst, lowest, mean, and current pain intensity, list current treatments and their perceived effectiveness, and judge the degree to which pain interferes with general activity, mood, walking ability, normal work, relationships with other individuals, sleep, and quality of life on a 10-point scale. This questionnaire is reliable and valid for use in persons with chronic low back pain.
The Brief Pain Inventory short form (BPI-sf) | day 7
  This nine-item questionnaire is used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. The patient is asked to rate the worst, lowest, mean, and current pain intensity, list current treatments and their perceived effectiveness, and judge the degree to which pain interferes with general activity, mood, walking ability, normal work, relationships with other individuals, sleep, and quality of life on a 10-point scale. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Modified Oswestry Disability Index (MODI) | Baseline
  This questionnaire evaluates the limitations individuals experience in their daily activities due to chronic low back pain. It consists of 10 items that can be scored on a 5-point scale. A percentage of restriction for the patient can be indicated on the basis of the total score. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Modified Oswestry Disability Index (MODI) | day 7
  This questionnaire evaluates the limitations individuals experience in their daily activities due to chronic low back pain. It consists of 10 items that can be scored on a 5-point scale. A percentage of restriction for the patient can be indicated on the basis of the total score. This questionnaire is reliable and valid for use in persons with chronic low back pain.
International Physical Activity Questionnaire short form (IPAQ) | Baseline
  This questionnaire is used to estimate physical activity level. The questionnaire consists of 7 questions. A higher score corresponds to a more physically demanding activity level. This questionnaire is reliable and valid for use in persons with chronic low back pain.
International Physical Activity Questionnaire short form (IPAQ) | day 7
  This questionnaire is used to estimate physical activity level. The questionnaire consists of 7 questions. A higher score corresponds to a more physically demanding activity level. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Depression Anxiety Stress Scale (DASS-21) | Baseline
  This scale was developed to examine depression, anxiety and stress without the major impact of possible somatic factors. The questions can be answered with 0 (not at all or never applicable), 1 (a little or sometimes applicable), 2 (quite or often applicable) or 3 (very definitely or mostly applicable). A qualification score of 1-5 (normal to very severe) is calculated for each scale. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Depression Anxiety Stress Scale (DASS-21) | day 7
  This scale was developed to examine depression, anxiety and stress without the major impact of possible somatic factors. The questions can be answered with 0 (not at all or never applicable), 1 (a little or sometimes applicable), 2 (quite or often applicable) or 3 (very definitely or mostly applicable). A qualification score of 1-5 (normal to very severe) is calculated for each scale. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Fear-Avoidance Components Scale (FACS) | baseline
  This questionnaire is designed to evaluate fear avoidance in patients with painful medical conditions and includes constructs such as pain-related catastrophic cognitions, hypervigilance, and avoidance behaviors. The FACS consists of 20 items with a score from 0 (totally disagree) to 5 (totally agree), with a total possible score of 100. The following anxiety avoidance severity levels are recommended for clinical interpretation: subclinical (0-20), mild (21-40), moderate (41-60), severe (61-80) and extreme (81-100) This questionnaire is reliable and valid for use in individuals with chronic low back pain.
Fear-Avoidance Components Scale (FACS) | day 7
  This questionnaire is designed to evaluate fear avoidance in patients with painful medical conditions and includes constructs such as pain-related catastrophic cognitions, hypervigilance, and avoidance behaviors. The FACS consists of 20 items with a score from 0 (totally disagree) to 5 (totally agree), with a total possible score of 100. The following anxiety avoidance severity levels are recommended for clinical interpretation: subclinical (0-20), mild (21-40), moderate (41-60), severe (61-80) and extreme (81-100) This questionnaire is reliable and valid for use in individuals with chronic low back pain.
Short form Health Survey (SF-36) | baseline
  This questionnaire provides an indication of the patient's multifactorial deficiencies by evaluating the general health status. It consists of 8 scores (vitality, physical functioning, physical pain, general perception of health, physical functioning in a role, emotional functioning in a role, social functioning in a role, mental health). The lower the score, the greater the dysfunction. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Short form Health Survey (SF-36) | day 7
  This questionnaire provides an indication of the patient's multifactorial deficiencies by evaluating the general health status. It consists of 8 scores (vitality, physical functioning, physical pain, general perception of health, physical functioning in a role, emotional functioning in a role, social functioning in a role, mental health). The lower the score, the greater the dysfunction. This questionnaire is reliable and valid for use in persons with chronic low back pain.
Pittsburg Sleep Quality Index (PSQI) | Baseline
  This validated questionnaire consisting of 19 questions evaluates last month's sleep quality grouped into 7 domains: sleep latency time, sleep duration, sleep medication, daytime functioning, sleep-related problems. Each domain is given a score from 0 to 3 and the global PSQI score ranges from 0 to 21. From a score> 5, one speaks of poor sleep quality.
Pittsburg Sleep Quality Index (PSQI) | day 7
  This validated questionnaire consisting of 19 questions evaluates last month's sleep quality grouped into 7 domains: sleep latency time, sleep duration, sleep medication, daytime functioning, sleep-related problems. Each domain is given a score from 0 to 3 and the global PSQI score ranges from 0 to 21. From a score> 5, one speaks of poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Annick Timmermanst, prof. dr., Principal Investigator — Hasselt University; Jonas Verbrugghe, dr., Study Chair — Hasselt University
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium

REFERENCES:
- [Background] McBeth J, Jones K. Epidemiology of chronic musculoskeletal pain. Best Pract Res Clin Rheumatol. 2007 Jun;21(3):403-25. doi: 10.1016/j.berh.2007.03.003. PMID 17602991
- [Background] Cimmino MA, Ferrone C, Cutolo M. Epidemiology of chronic musculoskeletal pain. Best Pract Res Clin Rheumatol. 2011 Apr;25(2):173-83. doi: 10.1016/j.berh.2010.01.012. PMID 22094194
- [Background] Woolf AD, Erwin J, March L. The need to address the burden of musculoskeletal conditions. Best Pract Res Clin Rheumatol. 2012 Apr;26(2):183-224. doi: 10.1016/j.berh.2012.03.005. PMID 22794094
- [Background] March L, Smith EU, Hoy DG, Cross MJ, Sanchez-Riera L, Blyth F, Buchbinder R, Vos T, Woolf AD. Burden of disability due to musculoskeletal (MSK) disorders. Best Pract Res Clin Rheumatol. 2014 Jun;28(3):353-66. doi: 10.1016/j.berh.2014.08.002. Epub 2014 Nov 18. PMID 25481420
- [Background] Moore, G., Durstine, J. L., Painter, P., & American College of Sports Medicine. (2016). Acsm's exercise management for persons with chronic diseases and disabilities, 4E. Human Kinetics.
- [Background] Manley, A. F. (1996). Physical activity and health: A report of the Surgeon General.
- [Background] Booth J, Moseley GL, Schiltenwolf M, Cashin A, Davies M, Hubscher M. Exercise for chronic musculoskeletal pain: A biopsychosocial approach. Musculoskeletal Care. 2017 Dec;15(4):413-421. doi: 10.1002/msc.1191. Epub 2017 Mar 30. PMID 28371175
- [Background] Smith BE, Hendrick P, Bateman M, Holden S, Littlewood C, Smith TO, Logan P. Musculoskeletal pain and exercise-challenging existing paradigms and introducing new. Br J Sports Med. 2019 Jul;53(14):907-912. doi: 10.1136/bjsports-2017-098983. Epub 2018 Jun 20. No abstract available. PMID 29925503
- [Background] Wilson, F., Gormley, J., & Hussey, J. (Eds.). (2011). Exercise therapy in the management of musculoskeletal disorders. Wiley-Blackwell.
- [Background] O'Riordan C, Clifford A, Van De Ven P, Nelson J. Chronic neck pain and exercise interventions: frequency, intensity, time, and type principle. Arch Phys Med Rehabil. 2014 Apr;95(4):770-83. doi: 10.1016/j.apmr.2013.11.015. Epub 2013 Dec 12. PMID 24333741
- [Background] Hunter DJ, Eckstein F. Exercise and osteoarthritis. J Anat. 2009 Feb;214(2):197-207. doi: 10.1111/j.1469-7580.2008.01013.x. PMID 19207981
- [Background] Fink, L., & Lewis, D. (2017). Exercise as a treatment for fibromyalgia: a scoping review. The Journal for Nurse Practitioners, 13(8), 546-551.
- [Background] Searle A, Spink M, Ho A, Chuter V. Exercise interventions for the treatment of chronic low back pain: a systematic review and meta-analysis of randomised controlled trials. Clin Rehabil. 2015 Dec;29(12):1155-67. doi: 10.1177/0269215515570379. Epub 2015 Feb 13. PMID 25681408
- [Background] Lima LV, Abner TSS, Sluka KA. Does exercise increase or decrease pain? Central mechanisms underlying these two phenomena. J Physiol. 2017 Jul 1;595(13):4141-4150. doi: 10.1113/JP273355. Epub 2017 May 26. PMID 28369946
- [Background] Rice D, Nijs J, Kosek E, Wideman T, Hasenbring MI, Koltyn K, Graven-Nielsen T, Polli A. Exercise-Induced Hypoalgesia in Pain-Free and Chronic Pain Populations: State of the Art and Future Directions. J Pain. 2019 Nov;20(11):1249-1266. doi: 10.1016/j.jpain.2019.03.005. Epub 2019 Mar 21. PMID 30904519
- [Background] Naugle KM, Fillingim RB, Riley JL 3rd. A meta-analytic review of the hypoalgesic effects of exercise. J Pain. 2012 Dec;13(12):1139-50. doi: 10.1016/j.jpain.2012.09.006. Epub 2012 Nov 8. PMID 23141188
- [Background] Naugle KM, Naugle KE, Fillingim RB, Samuels B, Riley JL 3rd. Intensity thresholds for aerobic exercise-induced hypoalgesia. Med Sci Sports Exerc. 2014 Apr;46(4):817-25. doi: 10.1249/MSS.0000000000000143. PMID 24002342
- [Background] Polaski AM, Phelps AL, Kostek MC, Szucs KA, Kolber BJ. Exercise-induced hypoalgesia: A meta-analysis of exercise dosing for the treatment of chronic pain. PLoS One. 2019 Jan 9;14(1):e0210418. doi: 10.1371/journal.pone.0210418. eCollection 2019. PMID 30625201
- [Background] Georgopoulos V, Akin-Akinyosoye K, Zhang W, McWilliams DF, Hendrick P, Walsh DA. Quantitative sensory testing and predicting outcomes for musculoskeletal pain, disability, and negative affect: a systematic review and meta-analysis. Pain. 2019 Sep;160(9):1920-1932. doi: 10.1097/j.pain.0000000000001590. PMID 31045746
- [Background] Kuithan P, Heneghan NR, Rushton A, Sanderson A, Falla D. Lack of Exercise-Induced Hypoalgesia to Repetitive Back Movement in People with Chronic Low Back Pain. Pain Pract. 2019 Sep;19(7):740-750. doi: 10.1111/papr.12804. Epub 2019 Jul 7. PMID 31187932
- [Background] van den Berg R, Jongbloed EM, de Schepper EIT, Bierma-Zeinstra SMA, Koes BW, Luijsterburg PAJ. The association between pro-inflammatory biomarkers and nonspecific low back pain: a systematic review. Spine J. 2018 Nov;18(11):2140-2151. doi: 10.1016/j.spinee.2018.06.349. Epub 2018 Jun 28. PMID 29960111
- [Background] Kawi J, Lukkahatai N, Inouye J, Thomason D, Connelly K. Effects of Exercise on Select Biomarkers and Associated Outcomes in Chronic Pain Conditions: Systematic Review. Biol Res Nurs. 2016 Mar;18(2):147-59. doi: 10.1177/1099800415599252. Epub 2015 Aug 14. PMID 26276511
- [Background] Svensson CI. Interleukin-6: a local pain trigger? Arthritis Res Ther. 2010;12(5):145. doi: 10.1186/ar3138. Epub 2010 Oct 28. PMID 21067533
- [Background] Zhou YQ, Liu Z, Liu ZH, Chen SP, Li M, Shahveranov A, Ye DW, Tian YK. Interleukin-6: an emerging regulator of pathological pain. J Neuroinflammation. 2016 Jun 7;13(1):141. doi: 10.1186/s12974-016-0607-6. PMID 27267059
- [Background] Munneke W, Ickmans K, Voogt L. The Association of Psychosocial Factors and Exercise-Induced Hypoalgesia in Healthy People and People With Musculoskeletal Pain: A Systematic Review. Pain Pract. 2020 Jul;20(6):676-694. doi: 10.1111/papr.12894. Epub 2020 May 15. PMID 32255268
- [Background] Lazaridou A, Martel MO, Cahalan CM, Cornelius MC, Franceschelli O, Campbell CM, Haythornthwaite JA, Smith M, Riley J, Edwards RR. The impact of anxiety and catastrophizing on interleukin-6 responses to acute painful stress. J Pain Res. 2018 Mar 28;11:637-647. doi: 10.2147/JPR.S147735. eCollection 2018. PMID 29636630
- [Background] Heffner KL, France CR, Trost Z, Ng HM, Pigeon WR. Chronic low back pain, sleep disturbance, and interleukin-6. Clin J Pain. 2011 Jan;27(1):35-41. doi: 10.1097/ajp.0b013e3181eef761. PMID 21188850
- [Background] Vaegter HB, Hoeger Bement M, Madsen AB, Fridriksson J, Dasa M, Graven-Nielsen T. Exercise increases pressure pain tolerance but not pressure and heat pain thresholds in healthy young men. Eur J Pain. 2017 Jan;21(1):73-81. doi: 10.1002/ejp.901. Epub 2016 Jun 5. PMID 27264211
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] Graven-Nielsen T, Vaegter HB, Finocchietti S, Handberg G, Arendt-Nielsen L. Assessment of musculoskeletal pain sensitivity and temporal summation by cuff pressure algometry: a reliability study. Pain. 2015 Nov;156(11):2193-2202. doi: 10.1097/j.pain.0000000000000294. PMID 26172551